CLINICAL TRIAL: NCT06106464
Title: Acute Cardiometabolic Effects of Moderate-Intensity Aerobic Exercise Plus Interrupting Sitting With Different Frequencies of Low-Intensity Physical Activity-A Randomized Crossover Trial
Brief Title: Cardiometabolic Effects of Aerobic Exercise Plus Breaking Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasin Ak (Other)
Responsible Party: Sponsor-Investigator, Yasin Ak, Principal Investigator, Kastamonu University
Organization: Kastamonu University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LIPA Break
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Sedentary Behaviour; Sedentary Time
Keywords: sedentary break; prolonged sitting; blood lipids; blood pressure; aerobic exercise; walking
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise+6.5 h of prolonged sitting (Experimental): Participants will sit 6.5 hours after 30 minutes of moderate intensity aerobic exercise.
  Interventions: Other: Aerobic exercise+6.5 h of prolonged sitting
- Aerobic exercise+2 minutes of walking breaks every 30 minutes (Experimental): Participants will break prolonged sitting with 2 minutes of walking every 30 minutes after 30 minutes of moderate intensity aerobic exercise.
  Interventions: Other: Aerobic exercise+2 minutes of walking breaks every 30 minutes
- Aerobic exercise+4 minutes of walking breaks every 1-h (Experimental): Participants will break prolonged sitting with 4 minutes of walking every 1-h after 30 minutes of moderate intensity aerobic exercise.
  Interventions: Other: Aerobic exercise+4 minutes of walking breaks every 1-h
- Aerobic exercise+8 minutes of walking breaks every 2-h (Experimental): Participants will break prolonged sitting with 8 minutes of walking every 2-h after 30 minutes of moderate intensity aerobic exercise.
  Interventions: Other: Aerobic exercise+8 minutes of walking breaks every 2-h

INTERVENTIONS:
Other: Aerobic exercise+6.5 h of prolonged sitting — Volunteers, whose fasting blood samples are drawn and who eat a standard breakfast, will perform a 30-minute walking exercise on a treadmill at 40-45% of their heart rate reserve. They will then sit in the chair for 6.5 hours. While seated, volunteers will be asked not to leave their seats except to use the toilet. Volunteers will be able to read and use computers and phones while sitting. Venous and capillary blood samples will be drawn at regular intervals and their blood pressures will be measured.
  Arms: Aerobic exercise+6.5 h of prolonged sitting
Other: Aerobic exercise+2 minutes of walking breaks every 30 minutes — Volunteers, whose fasting blood samples are drawn and who eat a standard breakfast, will perform a 30-minute walking exercise on a treadmill at 40-45% of their heart rate reserve. They will then interrupt sitting with 2-minute walks at 35-40% of their heart rate reserve every 30 minutes for 6.5 hours after moderate-intensity aerobic exercise. They will make a twelve interruptions throughout 6.5 hours period and will have a total of 24 minutes of interruption throughout the intervention. While seated, volunteers will be asked not to leave their seats except to use the toilet. Volunteers will be able to read and use computers and phones while sitting. Venous and capillary blood samples will be drawn at regular intervals and their blood pressures will be measured.
  Arms: Aerobic exercise+2 minutes of walking breaks every 30 minutes
Other: Aerobic exercise+4 minutes of walking breaks every 1-h — Volunteers, whose fasting blood samples are drawn and who eat a standard breakfast, will perform a 30-minute walking exercise on a treadmill at 40-45% of their heart rate reserve. They will then interrupt sitting with 4-minute walks at 35-40% of their heart rate reserve every 1 hour for 6.5 hours after moderate-intensity aerobic exercise. They will make six interruptions throughout 6.5 hours period and will have a total of 24 minutes of interruption throughout the intervention. While seated, volunteers will be asked not to leave their seats except to use the toilet. Volunteers will be able to read and use computers and phones while sitting. Venous and capillary blood samples will be drawn at regular intervals and their blood pressures will be measured.
  Arms: Aerobic exercise+4 minutes of walking breaks every 1-h
Other: Aerobic exercise+8 minutes of walking breaks every 2-h — Volunteers, whose fasting blood samples are drawn and who eat a standard breakfast, will perform a 30-minute walking exercise on a treadmill at 40-45% of their heart rate reserve. They will then interrupt sitting with 8-minute walks at 35-40% of their heart rate reserve every 2 hour for 6.5 hours after moderate-intensity aerobic exercise. They will make six interruptions throughout 6.5 hours period and will have a total of 24 minutes of interruption throughout the intervention. While seated, volunteers will be asked not to leave their seats except to use the toilet. Volunteers will be able to read and use computers and phones while sitting. Venous and capillary blood samples will be drawn at regular intervals and their blood pressures will be measured.
  Arms: Aerobic exercise+8 minutes of walking breaks every 2-h

SUMMARY:
The goal of this randomized crossover clinical trial is to investigate the effects of interrupting prolonged sitting with intermittent walks of equal volume but at different frequencies, in addition to moderate-intensity aerobic exercise, on postprandial serum lipid profile in young adults between the ages of 18-30. The main questions it aims to answer are:

* Do interrupting prolonged sitting with intermittent walks of equal volume but at different frequencies sustain positive cardiometabolic effects after moderate-intensity aerobic exercise?
* If "yes", which frequency of breaks is more effective to provide cardiometabolic benefits?

Participants will complete four conditions on separate days: 1) 6.5 hours of prolonged sitting after 30 minutes of moderate intensity aerobic exercise 2) breaking prolonged sitting with 2 minutes of walking every 30 minutes after 30 minutes of moderate intensity exercise 3) breaking prolonged sitting with 4 minutes of walking every 1-h after 30 minutes of moderate intensity exercise 4) breaking prolonged sitting with 8 minutes of walking every 2-h after 30 minutes of moderate intensity aerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Being able to participate in physical activity
* More than 7 hours of daily sitting time measured subjectively
* Not exercising regularly in the last 3 months

Exclusion Criteria:

* Hypertension
* Coronary heart disease
* Heart failure
* Diabetes mellitus
* Metabolic syndrome
* Obesity
* Hypothyroidism
* Non-alcoholic fatty liver disease
* Chronic inflammatory joint disease
* Chronic renal failure
* Cushing's syndrome
* HIV infection
* Being on antihypertensive medication
* Being on lipid-lowering medication
* Being on antidiabetic medication
* Being on systemic glucocorticoid medication
* LDL-cholesterol≥130 mg.dL-1
* HDL-cholesterol <40 mg.dL-1 for men; <50 mg.dL-1 for women
* Prediabetes
* Alcohol addiction
* Smoking
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Capillary glucose area under the curve | During the four 7.5-hour intervention sessions samples will be collected at the 30th, 60th, 90th, 120th and 210th minutes after breakfast, and at the 30th, 60th, 90th, 120th and 210th minutes after lunch.
  Fasting and subsequent capillary blood glucose measurements will be carried out. Blood samples will be taken by pricking the tip of the distal phalanx of the right or left middle finger with a lancet. The first drop of blood will be wiped with cotton and the second drop of blood will be analyzed with a glucometer (GL 44, Beurer GmbH, Germany). Two consecutive measurements will be made and the average of both measurements will be recorded. For each 7.5-hour intervention, the total area under the curve (AUC) will be calculated for capillary glucose using the trapezoidal method. Incremental AUC will then be calculated by subtracting the area of baseline level from the total AUC.
Serum Low-Density Lipoprotein cholesterol area under the curve | During the four 7.5-hour intervention sessions, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch
  Fasting venous blood samples for serum LDL cholesterol will be collected by inserting a cannula into the appropriate vein. The intravenous cannula will be fixed tightly with patch tape. Then fasting blood samples will be drawn. During each 7.5-hour intervention, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch from the intravenous cannula with a syringe. The blood samples taken into the syringe will be transferred to a yellow capped gel tube and the blood samples will be sent to the biochemistry laboratory for analysis.For each 7.5-hour intervention, the total AUC will be calculated for serum LDL cholesterol using the trapezoidal method. Incremental AUC will then be calculated by subtracting the area of baseline level from the total AUC.
Serum High-Density Lipoprotein cholesterol area under the curve | During the four 7.5-hour intervention sessions, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch
  Fasting venous blood samples for serum HDL cholesterol will be collected by inserting a cannula into the appropriate vein. The intravenous cannula will be fixed tightly with patch tape. Then fasting blood samples will be drawn. During each 7.5-hour intervention, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch from the intravenous cannula with a syringe. The blood samples taken into the syringe will be transferred to a yellow capped gel tube and the blood samples will be sent to the biochemistry laboratory for analysis.For each 7.5-hour intervention, the total AUC will be calculated for serum HDL cholesterol using the trapezoidal method. Incremental AUC will then be calculated by subtracting the area of baseline level from the total AUC.
Serum total cholesterol area under the curve | During the four 7.5-hour intervention sessions, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch
  Fasting venous blood samples for serum total cholesterol will be collected by inserting a cannula into the appropriate vein. The intravenous cannula will be fixed tightly with patch tape. Then fasting blood samples will be drawn. During each 7.5-hour intervention, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch from the intravenous cannula with a syringe. The blood samples taken into the syringe will be transferred to a yellow capped gel tube and the blood samples will be sent to the biochemistry laboratory for analysis.For each 7.5-hour intervention, the total AUC will be calculated for serum total cholesterol using the trapezoidal method. Incremental AUC will then be calculated by subtracting the area of baseline level from the total AUC.
Serum triglycerides area under the curve | During the four 7.5-hour intervention sessions, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch
  Fasting venous blood samples for serum triglycerides will be collected by inserting a cannula into the appropriate vein. The intravenous cannula will be fixed tightly with patch tape. Then fasting blood samples will be drawn. During each 7.5-hour intervention, 5 mL blood samples will be drawn at the 60th, 120th and 210th minutes after breakfast and at the 60th, 120th and 210th minutes after lunch from the intravenous cannula with a syringe. The blood samples taken into the syringe will be transferred to a yellow capped gel tube and the blood samples will be sent to the biochemistry laboratory for analysis.For each 7.5-hour intervention, the total AUC will be calculated for serum triglycerides using the trapezoidal method. Incremental AUC will then be calculated by subtracting the area of baseline level from the total AUC.

SECONDARY OUTCOMES:
Systolic blood pressure | During the four 7.5-hour intervention sessions, measurements will be carried out approximately at the 20th minute of each hour (10:20, 11:20, 12:20, 13:20, 14:20, 15:20, 16:20)
  Systolic blood pressures will be measured in the arm in the morning before each intervention and at regular intervals during each intervention. Measurements will be taken in an upright position just before blood samples are taken and after a rest period of at least 10 minutes from the last exercise bout. Blood pressure measurements will be taken with a digital blood pressure monitor (BM 40, Beurer GmbH, Germany) in the arm. The first measurement will be taken at approximately 08:30 a.m and the next 7 measurements will be carried out approximately at the 20th minute of each hour (10:20, 11:20, 12:20, 13:20, 14:20, 15:20, 16:20). Three measurements will be made at one-minute intervals and the average value of the three measurements will be recorded.
Diastolic blood pressure | During the four 7.5-hour intervention sessions, measurements will be carried out approximately at the 20th minute of each hour (10:20, 11:20, 12:20, 13:20, 14:20, 15:20, 16:20)
  Diastolic blood pressures will be measured in the arm in the morning before each intervention and at regular intervals during each intervention. Measurements will be taken in an upright position just before blood samples are taken and after a rest period of at least 10 minutes from the last exercise bout. Blood pressure measurements will be taken with a digital blood pressure monitor (BM 40, Beurer GmbH, Germany) in the arm. The first measurement will be taken at approximately 08:30 a.m and the next 7 measurements will be carried out approximately at the 20th minute of each hour (10:20, 11:20, 12:20, 13:20, 14:20, 15:20, 16:20). Three measurements will be made at one-minute intervals and the average value of the three measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Çatalzeytin Vocational School, Kastamonu, Turkey (Türkiye)

REFERENCES:
- [Derived] Ak Y, Guzel Y, Akyel S, Tatar OD, Karabulut E, Karaca A. Hourly 4-minute walking breaks from sitting following aerobic exercise reduce postprandial non-HDL cholesterol in healthy young adults: A randomized crossover trial. J Clin Lipidol. 2025 May-Jun;19(3):638-648. doi: 10.1016/j.jacl.2025.03.007. Epub 2025 Mar 21. PMID 40246606